CLINICAL TRIAL: NCT07120568
Title: Clinical Charactaristics, Risk Factors and Outcomes of Stroke in Pediatric Patients at Assiut University Children's Hospital
Brief Title: Clinical Charactaristics , Risk Factors and Outcomes of Stroke in Pediatric Patients at Assiut University Children's Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Mamdouh, Resident doctor, Assiut University
Other Study IDs: AssiutU AUCH
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Summary of the study is to recognize clinical picture , to identify risk factors and evaluate outcomes of stroke in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

* All patients from 28 day till 18 years who will attend to neurology unit and neurology clinic at assiut University Children's Hospital during duration of the study,.

Exclusion Criteria:

* neonates
* patient older than 18 years
* patient not presented with stroke

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children prestented with neurological insult to neurology unit or neurology clinic
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1.recognize clinical picture of stroke in pediatrics 2.identfiy risk factors of stroke in pediatrics 3. evaluate outcomes of stroke in pediatrics | Start of October 2025 to the end of December 2026